CLINICAL TRIAL: NCT05294783
Title: The Single Leg Squat and Hold Test With Kinematic Analysis to Evaluate Dynamic Knee Stability in Patients With ACL Injury
Brief Title: The Single Leg Squat Test to Evaluate Dynamic Knee Stability After ACLR
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Xin He, Principal investigator, Chinese University of Hong Kong
Other Study IDs: 2018.134
Record Dates: First submitted 2022-03-10; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: ACL Injury
Keywords: single leg squat; knee instability; ACL reconstruction; Kinematics
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL injured patients: All the ACL injured patients recruited underwent ACL reconstruction with the same group of surgeons lead by the same chief surgeon.
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — ACL reconstruction is a standard surgery for ACL injured patients

SUMMARY:
Patients with anterior cruciate ligament (ACL) injury often suffer knee instability, which can be visualized as a wobbling knee during weight bearing exercises, such as the single leg squat. We propose to use the single-leg-squat-and-hold (SLSH) task with kinematic analysis to objectively evaluate dynamic knee stability in ACL injured patients. The aim of this study is (1) to compare knee kinematic variations capturing knee wobbling during SLSH between ACL subjects and healthy controls; and (2) to detect the changes in knee kinematic variations during SLSH following ACL reconstruction.

DETAILED DESCRIPTION:
Injuries to the anterior cruciate ligament (ACL) are common in pivoting sports such as soccer, handball, basketball and rugby. The ultimate goal of ACL reconstruction for most athletes is return-to-play. Despite successful surgery and a demanding rehabilitation process, some athletes still failed to return to play, and for those who returned to play, some would suffer a second ACL injury. With surgical reconstruction of the ACL, static knee stability can be restored, but dynamic knee stability may not . Patients with ACL injury often experience symptoms such as knee instability, feelings of "giving way" during activities. Biomechanically, dynamic knee stability is considered as the ability to control the relative tibiofemoral displacements during loading.

Regular monitoring of the knee stability before and after ACL reconstruction is necessary for medical personnel to design the most suitable rehabilitation program. In contrast to jumping and hopping tasks, squatting tasks present a similar weight bearing profile during knee flexion, but without the potentially risky landing phase. As poor knee dynamic knee stability can be visualized as a wobbling knee (frequent knee movements). In order to quantitatively and objectively evaluate dynamic knee stability from observing the knee wobbling motion, we propose a single leg squat and hold task(SLSH) with kinematic analysis. Kinematic curve derived from the SLSH involves both the magnitudes and the frequency of the motion fluctuation. This study aims (1) to compare knee kinematic variations capturing knee wobbling during SLSH between ACL-deficient patients who are scheduled for ACLR and healthy controls; and(2)to detect the changes in knee kinematic variations during SLSH following ACLR. We hypothesize that the ACL-deficient patients demonstrate greater knee kinematic variation than the healthy subjects and the knee kinematic variation will reduce after ACLR.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-35;
2. Participate in level I or level II sports with a Tegner score of more than 6 before injury(level I: sports involving jumping, cutting and pivoting, e.g.football, basketball etc; Level II: sports involving lateral movements, less pivoting than Level I eg. racket sports)
3. Scheduled for ACLR because of unilateral ACL injury;
4. Failure to meet any single criteria for a potential coper;
5. Contralateral knee without history of injury.

Exclusion Criteria:

1. Concomitant fracture, meniscus injury or full-thickness chondral injuries;
2. preoperative radiographic signs of arthritis;
3. Revision ACL surgery;
4. With ankle pain, hip pain, low back pain or spine pathology;
5. Woman with pregnancy.

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Elite or recreational athletes with ACL injury who suffer knee instability and require surgical reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline knee range of flexion-extension at 3 months after ACLR | three months post-operatively
  knee range of flexion-extension will be measured during 10s holding phase of the single leg squat and hold test
Changes from baseline knee range of varus-valgus at 3 months after ACLR | three months post-operatively
  knee range of virus-valgus will be measured during 10s holding phase of the single leg squat and hold test
Changes from baseline knee range of internal-external rotation at 3 months after ACLR | one month pre-operatively and three months post-operatively
  knee range of internal-external rotation will be measured during 10s holding phase of the single leg squat and hold test
Changes from baseline frequency of knee flexion-extension at 3 months after ACLR | three months post-operatively
  the frequency of the relative flexion-extension movements will be quantified by the number of peak appearances during 10s holding phase of the single leg squat and hold test
Changes from baseline frequency of knee varus-valgus at 3 months after ACLR | three months post-operatively
  the frequency of the relative varus-valgus movements will be quantified by the number of peak appearances during 10s holding phase of the single leg squat and hold test
Changes from baseline frequency of knee internal-external rotation | three months post-operatively
  he frequency of the relative internal-external movements will be quantified by the number of peak appearances during 10s holding phase of the single leg squat and hold test

SECONDARY OUTCOMES:
Changes from baseline International Knee Documentation Committee(IKDC) score at 3 months after ACLR | three months post-operatively
  The IKDC is consisted of 10 questions about symptoms and activity ranging from 0 to 100 where 100 implies perfect knee function

CONTACTS AND LOCATIONS:
Overall Officials: Xin HE, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No